CLINICAL TRIAL: NCT02456350
Title: Genetically Engineered T Cells Expressing an Anti-CD19 Chimeric Antigen Receptor for Treatment of Patients With B Cell Malignancies
Brief Title: Anti-CD19 Chimeric Antigen Receptor (CAR)-Transduced T Cell Therapy for Patients With B Cell Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Collaborators: Shenzhen Institute for Innovation and Translational Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201504001
Record Dates: First submitted 2015-05-12; First posted 2015-05-28 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Lymphocytic Leukemia; Acute Lymphocytic Leukemia; Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anti-CD19-CAR transduced T cells (Experimental): Patients will receive a lymphodepleting preconditioning regimen followed by anti-CD19- CAR-transduced T cells.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: Anti-CD19-CAR transduced T cells

INTERVENTIONS:
Drug: Fludarabine — On days -5 through -3, Fludarabine 30mg/m2 IV will be infused over 30 minutes.
Drug: Cyclophosphamide — On days -5 through -3, Cyclophosphamide 300mg/m2 IV will be infused over 60 minutes followed by fludarabine.
Biological: Anti-CD19-CAR transduced T cells — Modified cells will be infused IV over 30 minutes (2-4 days after the last dose of fludarabine).

SUMMARY:
Autologous T cells engineered to express an anti-CD19 chimeric antigen receptor (CAR) with a safety switch will be infused back to patients with B cell malignancies, including lymphoma and leukemia. The patients will be monitored after infusion of anti-CD19 CAR-transduced T cells for adverse events, persistence of anti-CD19 CAR-transduced T cells and treatment efficacy.

Objectives:

To evaluate the safety and the efficacy of anti-CD19 CAR-transduced T cell therapy for patients with B cell malignancies.

Eligibility:

Patients between 1 and 85 years of age, who have relapsed or refractory CD19-expressing B-cell malignancies (leukemia or lymphoma) that have not responded to standard treatments.

Patients with a history of allogeneic stem cell transplant who meet all eligibility criteria are eligible to participate.

Patients must have adequate organ functions.

Design:

* Peripheral blood from patients will be collected for isolation of peripheral blood mononuclear cells (PBMCs), which will be transduced with a lentiviral or retroviral vector encoding anti-CD19 CAR containing a CD28 and a CD3 zeta as costimulatory domains as well as a safety switch.
* Patients will receive a lymphodepleting preconditioning regimen to prepare their immune system to accept modified T cells.
* Patients will receive an infusion of their own modified T cells. They will remain in the hospital to be monitored for adverse events until they have recovered from the treatment.
* Patients will have frequent follow-up visits to monitor the persistence of modified T cells and efficacy of the treatment.

DETAILED DESCRIPTION:
Despite progress has been made to date in the treatment of patients with B cell malignancies, including leukemia and lymphoma, many patients with relapsed or refractory diseases do not respond to the standard treatments. It has been shown that anti-CD19 CAR-transduced T cells may be an effective approach to treat the relapsed or refractory diseases. The procedure involves collecting PBMCs from the patients and modifying the T cells to attack the malignant B cells. In this trial, autologous T cells engineered to express an anti-CD19 chimeric antigen receptor (CAR) containing the signaling domains of CD28 and CD3-zeta, and a safety switch will be infused back to patients with B cell malignancies, including lymphoma and leukemia. The patients will be pretreated with a lymphodepleting preconditioning regimen before the infusion of anti-CD19 CAR T cells, and will be monitored for adverse events, persistence of anti-CD19 CAR-transduced T cells and the treatment efficacy.

OBJECTIVES:

* Primary objectives
* To determine the safety and feasibility of the administration of anti-CD19 CAR transduced T cells in patients with CD19+ B-cell malignancies.
* Secondary objectives:
* To determine if the treatment regimen can result in clinical regression of B-cell malignancies in the patients as described above.
* To determine the in vivo persistency of the anti-CD19 CAR-transduced T cells.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a CD19+ B cell malignancy，including relapsed or refractory B cell leukemia and B cell lymphoma；
2. Patients with CD19+ B cell malignancies are not able to receive standard treatments and willing to participate in the trial.
3. Patients must have a measurable or evaluable disease at the time of enrollment, which may include any evidence of disease including minimal residual disease detected by flow cytometry, cytogenetics, or polymerase chain reaction (PCR) analysis；
4. patients are not eligible for autologous or allogeneic stem-cell transplantation (SCT) or relapsed after autologous or allogeneic stem-cell transplantation；
5. Patients with history of allogeneic stem cell transplantation are eligible, providing 6 months had elapsed from SCT, they have no evidence of active graft-versus-host disease and no longer taking immunosuppressive agents during the treatment.
6. Willing to sign a durable power of attorney；
7. Able to understand and sign the Informed Consent Document；
8. Performance status：ECOG 0-2；
9. Life expectancy：More than 3 months；
10. Patients of both genders must be willing to practice birth control for four months after receiving a lymphodepleting preconditioning regimen；
11. Female participants of reproductive potential must have a negative serum or urine pregnancy test performed within 48 hours before infusion, because of the potentially dangerous effects on the fetus；
12. There is no obvious dysfunctions in heart , liver and kidney, and the functions of vital organs are normal；
13. Serology： (1) Seronegative for HIV antibody； (2) Seronegative for hepatitis B virus (HBV) and hepatitis C virus (HCV).
14. Hematology： (1) Absolute neutrophil count ≥ 1000/mm3 without support of filgrastim； (2) Platelet count ≥ 50,000/mm3； (3) Hemoglobin > 8.0g/dL； (4) lymphocyte count ≤ 4000/mm3。
15. Chemistry： (1) AST and ALT ≤ 5 times upper limit of normal； (2) Serum creatinine ≤ 1.6 mg/dl； (3) Bilirubin ≤ 1.5 mg/dl（3.0 mg/dL in patients with Gilbert's syndrome）。
16. More than three weeks must have elapsed since any prior systemic therapy at the time of randomization, and patients' toxicities must have recovered to a grade 1 or less (except for alopecia or vitiligo)；
17. Normal cardiac ejection fraction and no evidence of pericardial effusion as determined by an echocardiogram；

18、More than 30 days must have elapsed since Monoclonal antibody therapy administered prior to apheresis.

Exclusion Criteria:

1. Patients that require urgent therapy due to tumor mass effects such as bowel obstruction or blood vessel compression；
2. Patients that have active hemolytic anemia；
3. Patients with detectable cerebrospinal fluid malignant cells or brain metastases or with a history of cerebrospinal fluid malignant cells or brain metastases, or any residual intracranial implants；
4. Women of child-bearing potential who are pregnant or breastfeeding；
5. Active systemic infections, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system；
6. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease)；
7. Concurrent opportunistic infections；
8. Concurrent Systemic steroid therapy；
9. History of severe immediate hypersensitivity reaction to any of the agents used in this study；
10. Patients with central nervous system (CNS) metastases or symptomatic CNS involvement (including cranial neuropathies or mass lesions)；
11. CNS-3 disease or traumatic spinal tap with POSITIVE Steinherz/Bleyer algorithm with cerebral spinal fluid involvement with malignancy will make any patient not eligible for this protocol；
12. Patients with cardiac atrial or cardiac ventricular lymphoma involvement；
13. Other anti-neoplastic investigational agents currently or within 30 days prior to start of the treatment；
14. Previous treatment with any gene therapy products.

Ages: 1 Year to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2015-04; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events | 8 weeks
  To evaluate the safety and feasibility of the administration of anti-CD19 CAR transduced T cells in patients with CD19+ B-cell malignancies.

SECONDARY OUTCOMES:
Number of participants with Clinical responses | 2 years
  To determine if the treatment regimen can result in clinical regression of B-cell malignancies in the patients as described above.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Second People's Hospital, The First Affiliated Hospital of Shenzhen University, Shenzhen, Guangdong, China

REFERENCES:
- [Derived] Zhou W, Chen W, Wan X, Luo C, Du X, Li X, Chen Q, Gao R, Zhang X, Xie M, Wang M. Benefits of Chimeric Antigen Receptor T-Cell Therapy for B-Cell Lymphoma. Front Genet. 2022 Jan 20;12:815679. doi: 10.3389/fgene.2021.815679. eCollection 2021. PMID 35126471